CLINICAL TRIAL: NCT01029756
Title: A Randomised Controlled Trial of Intubation by Inexperienced Anaesthetists, Comparing the The Pentax Airway Scope AWS-S100 Rigid Video Laryngoscope(Pentax AWS) and the Macintosh Laryngoscope.
Brief Title: Randomised Controlled Trial of Intubation, Comparing Pentax AWS Against Macintosh Laryngoscope.
Acronym: PAWS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Grampian (Other Government)
Collaborators: Research and Development Department, NHS Grampian (Unknown); University of Aberdeen (Other)
Responsible Party: Principal Investigator, Lewis Walker, Dr, NHS Grampian
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ARI PentaxAWS 10
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Anaesthesia; Airway Management; Videolaryngoscopy
Keywords: Pentax Airway Scope AWS S100; Pentax AWS; Macintosh; Laryngoscope; Video Laryngoscope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Macintosh Laryngoscope (Active Comparator)
  Interventions: Device: Macintosh Laryngoscope
- Pentax AWS Videolaryngoscope (Active Comparator)
  Interventions: Device: Pentax AWS Videolaryngoscope

INTERVENTIONS:
Device: Macintosh Laryngoscope — Device used to gain a direct view of the vocal cords, to enable an endotracheal tube to be passed into the trachea at induction of anaesthesia.
  Other Names: Direct laryngoscopy
  Arms: Macintosh Laryngoscope
Device: Pentax AWS Videolaryngoscope — Self-contained video laryngoscope with an integral colour-viewing screen mounted on the handle. A camera at the tip transmits an indirect image, which obviates the need to obtain a direct view of the vocal cords, when passing an endotracheal tube on induction of anaesthesia.
  Other Names: Videolaryngoscopy
  Arms: Pentax AWS Videolaryngoscope

SUMMARY:
A randomised controlled trial of intubation by inexperienced anaesthetists, comparing the The Pentax Airway Scope AWS-S100 Rigid Video Laryngoscope(Pentax AWS) and the Macintosh Laryngoscope.

DETAILED DESCRIPTION:
General anaesthesia often requires that the trachea be protected by intubation. This involves placement of a cuffed endotracheal tube into the trachea, after the onset of unconsciousness and muscle relaxation. Usually this requires the anaesthetist to obtain a direct view of the patient's vocal cords via the mouth, using a laryngoscope such as the Macintosh laryngoscope. The endotracheal tube is then guided through the vocal cords into the trachea.

Difficult or failed intubation, is a potentially serious and occasionally life threatening complication. This is the unexpected inability to place the endotracheal tube in the correct place. The commonest cause is a failure to achieve an adequate view of the vocal cords at laryngoscopy.

Failed or difficult intubation significantly delays establishment of a secure airway and therefore can lead to major morbidity from hypoxia and/or aspiration of gastric contents. Other morbidity can also ensue from delay to the procedure in emergency situations or airway trauma due the various devices used or the force required to secure intubation. Whilst all anaesthetists and their assistants are trained to deal with difficult or failed intubations, disasters do occur. For example, in obstetrics, the previous Confidential Enquiry into Maternal Deaths reported five of the six deaths directly due to anaesthesia were related to intubation difficulties.

The Pentax Airway Scope AWS-S100 (Pentax AWS), Rigid Video Laryngoscope for Intubation is a new self-contained video laryngoscope with an integral colour-viewing screen mounted on the handle. A camera at the tip transmits an indirect image, which obviates the need to obtain a direct view of the vocal cords. It requires no prior set-up of equipment and is intuitive to use for anyone already competent in traditional direct laryngoscopy. Previously conducted evaluations of the scope have been presented and show that intubation can be secured within a clinically normal time span by various grades of anaesthetists in various clinical situations. Authors are currently suggesting it has a role as a back-up device for difficult intubations and for training. One has been obtained for the Foresterhill site for these purposes.

RATIONALE The simplicity of use and intuitive function of the Pentax AWS suggests it may have a wider role than as a back-up and could possibly be the first-line laryngoscope for situations where difficulty with intubation is more likely or more hazardous.

The incidence of difficult or failed intubation for an individual anaesthetist is related to their experience, decreasing as experience increases.

The purpose of this trial is to evaluate the Pentax AWS when used by relatively inexperienced anaesthetists. Inexperienced anaesthetists are those most likely to encounter difficulties and thus their practice carries the highest risk. Therefore, this is a setting in which there would be a particular benefit to patient safety in having the most effective tool for successful and timely completion of tracheal intubation.

METHODS The study will compare intubation using the Pentax AWS vs. the usual Macintosh laryngoscope in a sample of patients where 1st and 2nd year specialist trainees in anaesthesia (ST's) perform the intubation. There will be no other change in routine practice for the purposes of the trial. Specifically, the trial will recruit only from the population of patients that the ST's are routinely scheduled to intubate anyway. They will be working under the direct supervision of a consultant or senior specialist registrar (SpR), at all times.

Initially, data relating to routine intubations with the Macintosh laryngoscope will be collected. We will conduct training in the method of use of the Pentax AWS with the ST's, to a pre-determined level (see below) and collect and compare learning data, during routine clinical work with this laryngoscope. Following on from this, we will determine the effectiveness of the Pentax AWS in patients undergoing routine tracheal intubation.

4 ST's will perform the intubations within the trial. They fulfil the experience criteria required of the study, they began anaesthetic training between August 2010 and August 2011, have reached the required Royal College of Anaesthetists' level of competency in the practice of intubation and are approved to anaesthetise with indirect supervision.

Prior to commencement of recruitment into this study, it will be necessary for these ST anaesthetists to demonstrate a safe level of ability with the Pentax AWS. This is in order not to compromise safety in those patients randomized to undergo intubation with the Pentax AWS. They will be trained in the use of the Pentax AWS by the principle investigator (PI), initially using an airway training manikin and then in normal clinical practice. After gaining basic skill with the Pentax AWS, intubation with this scope will be timed. Supervised training with the Pentax AWS will continue until the ST anaesthetist is able to intubate in a clinically safe timeframe and then ST anaesthetists will be required to perform this successfully without trainer input in ten consecutive procedures. Once assessed as competent with the Pentax AWS by the PI they will be eligible to intubate patients entering the trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and over)
* scheduled for elective surgery whose anaesthetic plan would normally include oral intubation using a Macintosh laryngoscope blade by a junior anaesthetist and who have given valid informed consent.

Exclusion Criteria:

* Patients requiring special techniques for intubation such as awake fibreoptic intubation.
* Unconscious or critically ill patients.
* Emergency situations.
* Vulnerable patients including patients with:

  * learning difficulties,
  * terminal illness, mental illness, dementia,
  * prisoners and
  * those who could be considered to have a particularly dependent relationship with the investigator(such as medical students).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Is there a clinically significant difference in the time taken to successfully intubate the trachea? | Following induction of anaesthesia

SECONDARY OUTCOMES:
Is there a difference in the Intubation Difficulty Score? | Measured at intubation

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Walker, MBChB,FRCA, Principal Investigator — Consultant Anaesthetist NHS Grampian
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, Grampian, United Kingdom